CLINICAL TRIAL: NCT05622786
Title: Effect of High-Intensity Gait Training Using a Treadmill on Locomotion Recovery in Traumatic Brain Injury Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment status
Sponsor: Carilion Clinic (Other)
Collaborators: Radford University (Other); Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Courtney Perkins, PT, DPT, Principal Investigator, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-21-1512
Record Dates: First submitted 2022-10-20; First posted 2022-11-21 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Traumatic Brain Injury; Gait Disorders, Neurologic
Keywords: High-intensity; Gait training; Traumatic Brain injury; Heart rate; Treadmill
MeSH Terms: conditions — Brain Injuries, Traumatic; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Treadmill Gait Training (HIGT) (Experimental): High-intensity walking physical therapy with some low intensity therapy.
  Interventions: Other: HIGT - physical rehab
- Low Intensity Physical Therapy (Active Comparator): Low-intensity gait activities, exercises (such as lower extremity strength training with or without weights or electrical stimulation, sit to stands from a chair, mat exercises for upper/lower extremities and core strength, etc.), stretches, balance training activities, and other therapeutic activities (such as transfers, bed mobility training, etc.).
  Interventions: Other: Low intensity physical therapy

INTERVENTIONS:
Other: HIGT - physical rehab — High Intensity Gait Training using treadmill and overhead harness for fall prevention
  Arms: High-Intensity Treadmill Gait Training (HIGT)
Other: Low intensity physical therapy — Low Intensity Gait Activities
  Arms: Low Intensity Physical Therapy

SUMMARY:
The project will consist of subjects who have suffered Traumatic Brain Injury (TBI) and who are able to ambulate on treadmill with or without a harness system. This will be a 4-week controlled study consisting of two groups of TBI patients, high-intensity intervention group and low-intensity control group. Both groups will receive physical therapy treatment 3 times per week for 1 hour. The intervention group will undergo 30-minute sessions of high-intensity walking on a treadmill with an overhead harness attached for safety. In addition, they will also get up to 30-minutes of low-intensity physical therapy in order to receive 1 hour of treatment time. The control group will undergo only low-intensity physical therapy activities for 1-hour. Low-intensity physical therapy will include strength exercises, stretches, balance, and low-intensity gait training. All participants in both groups will complete these outcome measures on the first day of the study, after 2 weeks of participation, and again at the end of 4 weeks or on their last day before discharge from Carilion's services. Later on, all participants in both groups will be followed up to complete the same set of outcome measures at the end of 1 month since completion of the protocol. This follow up session will take up to 45 minutes to complete.

DETAILED DESCRIPTION:
Gait, mobility and cognitive function will be first assessed using seven standardized performance-based outcome measures including both mobility and cognitive measures. All participants in both groups will complete these outcome measures on the first day of the study, after 2 weeks of participation, again at the end of 4 weeks, or on their last day before being discharged from Carilion's services, and 1 month after their 4 week completion.

Participants of the intervention group will undergo physical therapy for 3 days a week for 4 weeks, with each session lasting a total of 60 minutes. They will start with 30 minutes of high-intensity gait training (HIGT) followed by up to 30 minutes of low-intensity therapy. For HIGT, participants will be secured safely on a treadmill with or without an overhead harness and unweighting system for successful gait training. Their resting HR and BP would be noted. Participants would begin with a warmup for 3 minutes by walking at low speeds with intensity of 30-50% of heart rate reserve (HRR). HR would be monitored continuously from here onwards till the conclusion of the protocol. Following the warmup, treadmill walking speed will be initially set at target HR of 85%HRR that was noted from the treadmill test. If the participant did not reach 85% HRR during the treadmill test, treadmill speed would be set by subtracting 0.1 mph (or 0.1 treadmill workload unit) from the speed at which they started showing gait instability or backward drift during the treadmill test. The goal would be to have participants walk at high aerobic intensity with target HR between 60-85%HRR, ideally close to 85%HRR, for 25 minutes. The studies report that the closer the heart rate can be maintained to the 85% target HR, the more beneficial the training.

If a participant is unable to achieve at least 60%HRR in the first few minutes of high-intensity phase, the participant's feeling of physical exertion would also be measured by asking them about a score on the Rates of Perceived Exertion (RPE) scale of 0-10. Here the goal would be to have them maintain an exertion intensity score of 5-8. If needed, participants would be allowed to rest by standing or sitting down. The amount of time spent in high-intensity and rest periods would be recorded. BP will also be recorded at 15-minute and 25-minute timepoints, or during rest breaks. At conclusion of 25 minutes of HIGT, participants will cool down for 2 minutes by walking at 30-50% HRR. Their HR and BP will again be measured at the end of the cool down period. Besides HR and BP, participant's oxygen saturation would also be monitored during this protocol using a pulse oximeter to assess blood oxygen levels. Depending on the remaining time and activity tolerance levels, intervention group participants will then perform up to 30 minutes of low-intensity physical therapy until they have reached a total of 60 minutes for that session. These may consist of low-intensity gait activities, exercises (such as lower extremity strength training with or without weights or electrical stimulation, sit to stands from a chair, mat exercises for upper/lower extremities and core strength, etc.), stretches, balance, and other therapeutic activities (such as transfers, bed mobility training, etc.) for functional mobility.

Participants in the control group will receive 60-minute sessions of only low-intensity physical therapy for 3 days a week for 4 weeks. Here, the goal is to have the participants work at a lower intensity with a target HR below 60%HRR. Low-intensity physical therapy could include low-intensity gait activities, exercises (such as lower extremity strength training with or without weights or electrical stimulation, sit to stands from a chair, mat exercises for upper/lower extremities and core strength, etc.), stretches, balance, and other therapeutic activities (such as transfers, bed mobility training, etc.). During these sessions, HR and BP would be measured and noted at regular intervals to monitor and note the cardiorespiratory intensity of those activities.

ELIGIBILITY:
Inclusion Criteria:

* Medical and treadmill screening clearance to participate in this study
* Persons with mild, moderate, or severe Traumatic Brain Injury at onset (first time or repeats)
* 18-65 years old persons who are able to ambulate on treadmill with or without assistive devices and with or without need for bodyweight-support harness system
* Ability to communicate with investigators to follow protocol instructions and respond appropriately
* Patients who have decision-making capacity and are able to consent for themselves

Exclusion Criteria:

* Unstable orthopedic conditions, for example, unstable craniectomies or weight-bearing restrictions.
* Unstable cardiac conditions including, unstable angina, unstable cardiac dysrhythmias, myocardial ischemia or hypertension at rest (systolic BP > 140mm Hg and diastolic BP >90 mm Hg, or if over this range, then a physician must clear patient for participation)
* Acute systemic infection accompanied by fever, body aches or swollen lymph glands.
* Hospitalization for acute cardiac, pulmonary or metabolic conditions in the past 3 months.
* Any other physical or mental restrictions preventing participation in the research protocol.
* Women who are pregnant are being excluded as this is considered a high risk study. They will be asked via verbal questioning via the following statements, "Are you currently pregnant?" or "Are you planning to become pregnant?".
* Non-English Speakers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Five Times Sit to Stand Test | Through intervention and follow-up period, up to 8 weeks. This would be administered at the beginning, at the end of 2 weeks, at the end of 4 weeks of interventions, and finally at the end of 4 weeks following end of interventions for follow-up.
  Stand up and sit down as quickly as possible 5 times, keeping your arms folded across your chest.
Six Minute Walk Test (6MWT) | Through intervention and follow-up period, up to 8 weeks. This would be administered at the beginning, at the end of 2 weeks, at the end of 4 weeks of interventions, and finally at the end of 4 weeks following end of interventions for follow-up.
  a sub-maximal exercise test used to assess walking endurance and aerobic capacity. Participants will walk around the perimeter of a set circuit for a total of six minutes.
10 Meter Walk Test (10mWT) | Through intervention and follow-up period, up to 8 weeks. This would be administered at the beginning, at the end of 2 weeks, at the end of 4 weeks of interventions, and finally at the end of 4 weeks following end of interventions for follow-up.
  Assesses walking speed in meters/second (m/s) over a short distance.
Berg Balance Scale (BBS) | Through intervention and follow-up period, up to 8 weeks. This would be administered at the beginning, at the end of 2 weeks, at the end of 4 weeks of interventions, and finally at the end of 4 weeks following end of interventions for follow-up.
  Used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. The minimum value of this assessment is 0, and the maximum is 56. A higher score means a better outcome.
Timed Up and Go (TUG) | Through intervention and follow-up period, up to 8 weeks. This would be administered at the beginning, at the end of 2 weeks, at the end of 4 weeks of interventions, and finally at the end of 4 weeks following end of interventions for follow-up.
  Assesses a person's mobility that requires both static and dynamic balance.
Timed Up and Go (Cognitive) | Through intervention and follow-up period, up to 8 weeks. This would be administered at the beginning, at the end of 2 weeks, at the end of 4 weeks of interventions, and finally at the end of 4 weeks following end of interventions for follow-up.
  Complete a TUG test while counting backward by three from a randomly selected number between 20 and 100.
Montreal Cognitive Assessment (MoCA) | Through intervention and follow-up period, up to 8 weeks. This would be administered at the beginning, at the end of 2 weeks, at the end of 4 weeks of interventions, and finally at the end of 4 weeks following end of interventions for follow-up.
  A rapid screening instrument for mild cognitive dysfunction. The minimum value of this assessment is 0, and the maximum is 30. A higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Perkins, DPT, Principal Investigator — Carilion Clinic
Locations (1):
- Institute for Orthopaedics and Neurosciences, Roanoke, Virginia, United States

REFERENCES:
- [Result] Hornby TG, Reisman DS, Ward IG, Scheets PL, Miller A, Haddad D, Fox EJ, Fritz NE, Hawkins K, Henderson CE, Hendron KL, Holleran CL, Lynskey JE, Walter A; and the Locomotor CPG Appraisal Team. Clinical Practice Guideline to Improve Locomotor Function Following Chronic Stroke, Incomplete Spinal Cord Injury, and Brain Injury. J Neurol Phys Ther. 2020 Jan;44(1):49-100. doi: 10.1097/NPT.0000000000000303. PMID 31834165
- [Result] Moore JL, Nordvik JE, Erichsen A, Rosseland I, Bo E, Hornby TG; FIRST-Oslo Team. Implementation of High-Intensity Stepping Training During Inpatient Stroke Rehabilitation Improves Functional Outcomes. Stroke. 2020 Feb;51(2):563-570. doi: 10.1161/STROKEAHA.119.027450. Epub 2019 Dec 30. PMID 31884902
- [Result] Holleran CL, Rodriguez KS, Echauz A, Leech KA, Hornby TG. Potential contributions of training intensity on locomotor performance in individuals with chronic stroke. J Neurol Phys Ther. 2015 Apr;39(2):95-102. doi: 10.1097/NPT.0000000000000077. PMID 25784587
- [Result] Ada L, Dean CM, Morris ME, Simpson JM, Katrak P. Randomized trial of treadmill walking with body weight support to establish walking in subacute stroke: the MOBILISE trial. Stroke. 2010 Jun;41(6):1237-42. doi: 10.1161/STROKEAHA.109.569483. Epub 2010 Apr 22. PMID 20413741
- [Result] Macko RF, Ivey FM, Forrester LW, Hanley D, Sorkin JD, Katzel LI, Silver KH, Goldberg AP. Treadmill exercise rehabilitation improves ambulatory function and cardiovascular fitness in patients with chronic stroke: a randomized, controlled trial. Stroke. 2005 Oct;36(10):2206-11. doi: 10.1161/01.STR.0000181076.91805.89. Epub 2005 Sep 8. PMID 16151035
- [Result] Holleran CL, Hennessey PW, Leddy AL, Mahtani GB, Brazg G, Schmit BD, Hornby TG. High-Intensity Variable Stepping Training in Patients With Motor Incomplete Spinal Cord Injury: A Case Series. J Neurol Phys Ther. 2018 Apr;42(2):94-101. doi: 10.1097/NPT.0000000000000217. PMID 29547484
- [Result] Ardestani MM, Henderson CE, Salehi SH, Mahtani GB, Schmit BD, Hornby TG. Kinematic and Neuromuscular Adaptations in Incomplete Spinal Cord Injury after High- versus Low-Intensity Locomotor Training. J Neurotrauma. 2019 Jun 15;36(12):2036-2044. doi: 10.1089/neu.2018.5900. Epub 2019 Feb 1. PMID 30362878
- [Result] Gadelha A, Voigtmann C. High Intensity Gait Training in Anoxic Brain Injury: A Case Study. Archives of Physical Medicine and Rehabilitation. DOE: https://doi.org/10.1016/j.apmr.2021.07.596

DOCUMENTS (1):
  • Informed Consent Form (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT05622786/ICF_000.pdf